CLINICAL TRIAL: NCT02296879
Title: A Multicenter, Open Label, Phase I Dose Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Intravenous SAIT301 in Subjects With Advanced c-MET Positive (+) Solid Tumors Followed by Expansion in Selected Tumor Types
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Young Suk Park (Other)
Responsible Party: Sponsor-Investigator, Young Suk Park, Samsung Medical Center, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-09-077
Record Dates: First submitted 2014-11-18; First posted 2014-11-20 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Solid Tumors
MeSH Terms: interventions — SAIT301

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SAIT301 (Experimental): For Stage 1, subjects will be sequentially assigned to 1 of approximately 8 cohorts comprised of 3 to 6 subjects each. SAIT301 will be administered according to a modified Fibonacci sequence and following a 3 + 3 design.
  For Stage 2, the MTD or (RP2D) determined in the Stage 1 will be administered to additional subjects with selected diagnoses, 15 subjects per selected diagnosis. After completion of Stage 1 the SRC may elect to increase the interval between doses (i.e., increase cycle length to 28 days) based on the emerging PK data from the lower SAIT301 dose levels.
  Interventions: Genetic: SAIT301

INTERVENTIONS:
Genetic: SAIT301 — The treatment period will consist of 21-day cycles. On Day 1 of each cycle, SAIT301 will be administered as an intravenous (IV) infusion.

SUMMARY:
Mesenchymal epithelial transition factor (c-MET) is a receptor tyrosine kinase that, when engaged by its ligand hepatocyte growth factor (HGF), has been implicated in various cellular process including development as well as oncogenesis.

SAIT301 is a novel humanized monoclonal antibody targeting the alpha chain of extracellular domain of c-MET. Binding of SAIT301 to c-MET blocks HGF binding and inhibits HGF-mediated signaling. Furthermore, SAIT301 also induces efficient c-MET internalization from the cell surface and subsequent degradation, resulting in inhibition of growth of the c-MET addicted cancer cells.

The sponsor decided to enroll subjects with tumors that express c-MET (by immunohistochemistry [IHC]) for this study, as the subjects with no c-MET expression are unlikely to benefit from SAIT301 treatment.

Stage 1 of this Phase I study is designed to evaluate the safety, tolerability, pharmacokinetic (PK) profile, and anti-tumor activity of SAIT301 administered as a single IV infusion in 21 day cycles, for up to 4 cycles. Subjects without evidence of tumor progression after 4 cycles will be eligible to continue on SAIT301 treatment if there is no evidence of tumor progression for a further 4 cycles (Cycles 5 to 8). Biomarkers related to SAIT301 and/or tumor response will also be evaluated.Stage 2 will further evaluate the safety and PK profile of SAIT301 in select types of cancers. Dosing frequency may be adjusted based on the PK profile obtained during Stage 1.

DETAILED DESCRIPTION:
The primary objectives of the study are as follows:

* To evaluate the safety and tolerability of SAIT301.
* To determine the MTD of SAIT301 and the dose level of SAIT301 where dose limiting toxicity (DLT) is observed in subjects with advanced solid tumors or define recommended Phase II dose (RP2D) as an alternative to establishing the MTD.

Methodology: This first in man study will consist of 2 stages. Stage 1 will be a dose escalation study with a 3 + 3 design and will evaluate the safety, tolerability, PK profile, biomarkers, and preliminary anti-tumor activity of ascending doses of SAIT301 in subjects with c-MET + advanced solid tumors and define the MTD (or recommended Phase II dose [RP2D]) of SAIT301. If the PK trough levels exceed the minimum acceptable trough level for SAIT301 (25 μg/mL), the Safety Review Committee (SRC) may elect to terminate further dose escalation and declare a recommended Phase II dose (RP2D) and schedule as an alternative to establishing the MTD. In Stage 2 the MTD (or RP2D) defined in Stage 1 will be administered to additional subjects with selected diagnoses, 15 subjects per selected diagnosis, to further evaluate the safety and PK profile, and any evidence of anti tumor activity of SAIT301 in these populations. The tumor types to be included in Stage 2 will be defined in a protocol amendment at a time close to study execution based on information available at that time.

The treatment period will consist of 21-day cycles. On Day 1 of each cycle, SAIT301 will be administered as an intravenous (IV) infusion.

For dose level 1, the first subject will receive an IV infusion of SAIT301 on Cycle 1 Day 1 and will be followed for 21 days (Cycle 1).

If the first subject at dose level 1 experiences a DLT during Cycle 1, 1 additional subject will be enrolled and will receive dose level 1, which is 50% of dose level 1. If this subject at dose level -1 does not experience a DLT during Cycle 1, 2 more subjects will be enrolled at dose level -1.

If the first subject at dose level 1 does not experience a DLT during Cycle 1, the second and third subjects will receive SAIT301 at dose level 1 and will be followed for 21 days (Cycle 1). At the discretion of the SRC, if the first 3 subjects at dose level 1 do not experience a DLT during Cycle 1, dose level 2 may be administered in the next cohort. If one of these subjects experiences a DLT, the cohort will be expanded and evaluated as described below.

For dose level 2 and each subsequent dose level, 3 subjects will receive SAIT301 on Day 1 of Cycle 1 and will be followed for 21 days (Cycle 1). If none of the 3 subjects experience a DLT, the next dose level can be administered in the next cohort. If 1 or more of the first 3 subjects experience a DLT, 3 more subjects will receive the same dose level. Dose escalation will continue until at least 2 subjects in a cohort of 3 to 6 subjects experience a DLT (i.e., ≥33% of subjects with a DLT at that dose level). Considering the possibility of relatively low efficacy, each subjects of dose level 1 and 2 can be administered with higher dose level after their first administration. This individual dose escalation can be determined by Investigators when safety data of the higher dose level are available.

For both Stage 1 and 2, subjects will continue to receive the assigned dose level of SAIT301 until unacceptable toxicity, documented progression of disease, another criterion for discontinuation is met, or until 4 cycles have been completed.

Subjects without evidence of tumor progression after 4 cycles may continue on SAIT301 treatment if there is no evidence of tumor progression for a further 4 cycles (Cycles 5 to 8). Subjects without evidence of tumor progression at the completion of Cycle 8 will be eligible for a follow-on protocol.

Subjects who experience a DLT will be discontinued from further treatment. At the completion of the dose escalation stage, the SRC may for Stage 2 alter the dosing interval between cycles based on emerging PK data from lower SAIT301 dose levels.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older.
2. Have a histologically or cytologically confirmed advanced solid tumor that has recurred or progressed following standard therapy, or that has not responded to standard therapy, or for which there is no standard therapy, or the subject is not a candidate for standard therapy.
3. Tumor positive for c-MET expression as determined by IHC. Results should be available before the subject can proceed in the study.
4. Adequate tumor biopsy material should be available for IHC and fluorescence in situ hybridization (FISH) of c-MET and biomarker analysis at the time of enrollment (formalin-fixed, paraffin-embedded tumor block or 20 fresh cut unstained slides).
5. At least 28 days must have elapsed since the subject's prior systemic therapy, radiotherapy, or any major surgery (excluding diagnostic biopsy or venous access device placement). Surgery requiring local/epidural anesthesia must be completed at least 72 hours before the first administration of SAIT301. For concomitant medications with a known half-life of less than 36 hours (e.g., tyrosine kinase inhibitors), the duration of time since prior therapy can be reduced to 14 days provided any drug-related toxicities have resolved to Grade 1 or better. Hormonal therapy for prostate or breast cancer are allowed during the study.
6. For dose levels 1 to 3, subjects must, at a minimum, have evaluable disease according to RECIST 1.1 guidelines. For dose levels above level 3, subjects must have measureable disease (≥1 cm by spiral computerized tomography [CT] or ≥2 cm by standard CT).
7. An ECOG performance status of <2.
8. Life expectancy of >12 weeks, as judged by the investigator.
9. Female subjects must not be pregnant or breastfeeding, or at risk to become pregnant during the study. Fertile male and female subjects must agree to use an effective barrier method of birth control to avoid pregnancy from the time of providing informed consent until 90 days after the last administration of SAIT301.
10. Female subjects of childbearing potential must have a negative serum pregnancy test within 7 days of the first administration of SAIT301. For the purpose of this study, female subjects of childbearing potential are defined as all female subjects after puberty unless they are postmenopausal for at least 1 year, or are surgically sterile (hysterectomy or bilateral oophorectomy or tubal ligation).
11. Adequate organ function as indicated by the laboratory test results obtained within 7 days prior to the first administration of SAIT301:

    Hematologic: Absolute neutrophil count ≥1.5 x 109/L, platelet count ≥100 x 109/L, and hemoglobin ≥9.0 g/dL.

    Liver function: Serum bilirubin <2.0 mg/dL, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <3 x upper limit of normal (ULN) without liver involvement, or <5 x ULN with liver involvement.

    Renal: serum creatinine ≤1.5 mg/dL.
12. Willing and able to provide written informed consent and to comply with the protocol, visit schedule, and requirements.

Exclusion Criteria:

Subjects will not be entered in the study for any of the following reasons:

1. Received previous treatment with SAIT301 or a previous drug with c-MET inhibitory activity.
2. Received any chemotherapy, immunotherapy, vaccines, monoclonal antibodies, major surgery, or irradiation, whether conventional or investigational, within 28 days of the first administration of SAIT301 in this study.
3. History of prior allergic reactions to protein therapeutics.
4. Active, uncontrolled systemic infection considered opportunistic, life threatening, or clinically significant.
5. Symptomatic or untreated central nervous system metastases.
6. Not recovered from acute toxicity of any therapy received prior to enrollment.
7. Received systemic treatment for bacterial infection within 7 days of screening.
8. Positive test results for human immunodeficiency virus (HIV), hepatitis B (core immunoglobulin M antibody and/or surface antigen), or hepatitis C at screening.
9. Any other serious medical condition which in the investigator's opinion would preclude safe participation in the study.
10. Likely to be non-compliant or uncooperative during the study, as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-01-20 (Actual); Primary Completion 2017-03-15 (Actual); Study Completion 2017-06-20 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), adverse events (AEs) of at least Common Terminology Criteria for Adverse Events (CTCAE) Grade 3 severity, and discontinuations due to AEs. | Up to 25 weeks for each subject
  Adverse events will be evaluated and categorized in accordance with the CTCAE, version 4.03.
The maximum tolerated dose (MTD) of SAIT301 and the dose level of SAIT301 where dose limiting toxicity (DLT) is observed in subjects with advanced solid tumors | Up to 25 weeks for each subject
  The frequency of DLTs as part of the MTD determination process.
A recommended Phase II dose (RP2D) as an alternative to establishing the MTD. | Up to 25 weeks for each subject
  RP2D determination as an alternative to establishing the MTD

SECONDARY OUTCOMES:
The pharmacokinetic (PK) profile of SAIT301 | Up to 25 weeks for each subject
  Free SAIT301 for Cycle 1 and Cycle 4 over dosing observation period of 0 to 21 days: maximum observed serum concentration (Cmax), time to maximum serum concentration (tmax), area under the serum concentration-time curve from zero to the last quantifiable concentration (AUC0-t), area under the concentration-time curve over the dosing interval (AUC0-tau).
  Free SAIT301 for Cycle 1, if half-life can be estimated with acceptable accuracy and/or for Cycle 4 if data collected in Cycle 4 are representative of steady state: area under the serum concentration-time curve from zero extrapolated to infinity (AUC0-inf), elimination rate constant (λz), elimination half-life (t1/2), apparent clearance from serum (CL), and volume of distribution at steady-state (VSS).
Objective tumor response for target lesions based on Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1, as assessed by repeat computerized tomography (CT) or magnetic resonance imaging (MRI). | Up to 25 weeks for each subject
To assess the preliminary anti-tumor activity of SAIT301 when administered as a single agent in this subject population | Up to 25 weeks for each subject
  Development of anti-SAIT301 binding antibodies and neutralizing antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Park Yong Suk, MD,Ph.D., Principal Investigator — Samsung Medical Center,Seoul,Korea
Locations (1):
- Samsung Medical Center, Seoul, South Korea